CLINICAL TRIAL: NCT00509405
Title: Effect of Neutralization of Endogenous Acid Production on Bone Mineral Density and Microarchitectural Composition of Bone in Humans
Brief Title: Effect of Neutralization of Endogenous Acid Production on BMD and Bone Microarchitectural
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Principal Investigator, Reto Krapf, Professor of Medicine, Kantonsspital Baselland Bruderholz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 316/06; NFP 53: 4053-110259
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Endogenous acid production; metabolic acidosis; potassium citrate; osteoporosis; sarcopenia; hypertension; Effect of potassium citrate on bone mineral density and bone mass
MeSH Terms: conditions — Acidosis; Osteoporosis; Sarcopenia; Hypertension | interventions — Potassium Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Potassium citrate (Placebo Comparator)
  Interventions: Drug: potassium citrate

INTERVENTIONS:
Drug: potassium citrate — 6 times 10 mEq per day, oral for 24 months

SUMMARY:
Hypothesis: Neutralization of acid production induced by the Western diet with oral administration of potassium citrate increases bone mineral density and bone mass as well as skeletal muscle mass and strength in elderly people (> 65y).

DETAILED DESCRIPTION:
We will perform a prospective, randomized, placebo-controlled trial evaluating the effect of K citrate on bone mineral density, microarchitectural composition of bone,nutritional parameters, lean body mass, parameters of skeletal muscle mass and strength, 24h and exercise induced blood pressure changes in otherwise healthy, elderly ambulatory subjects of both genders.

Potassium citrate (60 mEq) is supplied as tablets with a wax matrix (10 mEq of citrate per tablet) and ingested in three doses/day. All subjects will receive daily oral 500 mg of calcium and 400 IU of vitamin D to ensure adequate calcium and vitamin D supply.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 65 to 80y, tscores at L2-L4 0 to -2.5

Exclusion Criteria:

* Treated or necessity to treat low BMD (t-score L2 to L4 <-2.5)
* Any major medical illness that would possibly need hospitalization and/or be followed by foreseeable complications within 12 months and/or have a life-expectancy of less than 5 years
* Stable serum creatinine > 150 umol/l and/or known Type IV renal-tubular acidosis (hyperkalemia)
* vegetarians
* concommitant drug prescriptions: systemic and topical glucocorticoids, systemically acting estrogens (topical allowed): both within the last 6 months. antiosteoporosis drugs: bisphosphoponates, fluoride, calcitonin, all within the previous 12 months.
* vitamin D deficiency at screening visit
* technical difficulties to delineate bone area of interest during the screening visit

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 202 (Actual)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
BMD at L2-L4 by DEXA and microarchitectural composition of bone in both tibias and radius | 12 and 24 months

SECONDARY OUTCOMES:
Effect on BMD at hip and total body Effect on 24h ambulatory blood pressure | 12 and 24 months
effect on skeletal muscle mass and strength | 12 and 24 months
effect on left ventricular muscle mass | 24 months
effect on carotid media-intima thickness | 24 months
Hypoxia-induced endothelial vasorelaxation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Reto Krapf, MD, Principal Investigator — Department of Medicine, Kantonsspital Bruderholz, CH-4101 Bruderholz/Switzerland
Locations (1):
- Department of Medicine, Kantonsspital Bruderholz, Bruderholz/Basel, Basel-Landschaft, Switzerland

REFERENCES:
- See also: check in archive for "essen wir zu sauer" — http://www.medicalforum.ch